CLINICAL TRIAL: NCT06437509
Title: A Phase II Clinical Trial to Evaluate the Efficacy and Safety of BL-B01D1+PD-1 Monoclonal Antibody in Patients With Extensive-stage Small Cell Lung Cancer
Brief Title: A Study of BL-B01D1+PD-1 Monoclonal Antibody in Patients With Extensive-stage Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-B01D1-204-01
Record Dates: First submitted 2024-05-27; First posted 2024-05-31 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Extensive-stage Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study treatment (Experimental): Participants receive BL-B01D1 + PD-1 monoclonal antibody as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-B01D1; Drug: PD-1 monoclonal antibody

INTERVENTIONS:
Drug: BL-B01D1 — Administration by intravenous infusion for a cycle of 3 weeks.
  Other Names: iza-bren; izalontamab brengitecan; BMS-986507
Drug: PD-1 monoclonal antibody — Administration by intravenous infusion for a cycle of 3 weeks.

SUMMARY:
This study is a phase II clinical study to explore the efficacy and safety of BL-B01D1 + PD-1 monoclonal antibody combination therapy in patients with extensive-stage small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Subject volunteered to participate in the study and signed an informed consent;
2. Male or female aged ≥18 years and ≤75 years;
3. Expected survival time ≥3 months;
4. ECOG score 0-1;
5. Newly diagnosed patients with extensive-stage small cell lung cancer confirmed by histopathology and / or cytology;
6. A archived tumor tissue sample or fresh tissue sample of the primary or metastatic lesion must be provided within 3 years;
7. At least one measurable lesion meeting the RECIST v1.1 definition was required;
8. No blood transfusion and no use of cell growth factors and/or platelet-raising drugs within 14 days before screening, and the organ function level must meet the requirements;
9. The toxicity of previous antineoplastic therapy has returned to ≤ grade 1 as defined by NCI-CTCAE v5.0;
10. For premenopausal women of childbearing potential, a pregnancy test must be performed within 7 days before the initiation of treatment, a serum or urine pregnancy test must be negative, and the patient must not be lactating; All enrolled patients should take adequate barrier contraception during the entire treatment cycle and for 6 months after the end of treatment.

Exclusion Criteria:

1. Prior use of ADC drug therapy with small molecule toxins as topoisomerase I inhibitors;
2. Prior treatment with any systemic anti-tumor regimen for extensive-stage small cell lung cancer;
3. Pathology suggested small cell carcinoma containing non-small cell carcinoma components;
4. Subjects had used immunomodulatory drugs within 14 days before the first use of the study drug ;
5. Screening the history of severe cardiovascular and cerebrovascular diseases in the first half of the year ;
6. QT interval prolongation, complete left bundle branch block, III degree atrioventricular block, frequent and uncontrollable arrhythmia ;
7. Active autoimmune diseases and inflammatory diseases ;
8. Receiving long-term systemic corticosteroid therapy or equivalent anti-inflammatory active drugs or any form of immunosuppressive therapy prior to the first dose;
9. Other malignancies that have progressed or require treatment within 5 years prior to the first dose;
10. Have ILD requiring steroid therapy, or currently have ILD, or suspected ILD at screening;
11. Prior to initiation of study treatment, there were: a) poorly controlled diabetes mellitus; b) with severe complications of diabetes; c) glycosylated hemoglobin levels of 8% or more; d) hypertension that is poorly controlled by two antihypertensive drugs; e) history of hypertensive crisis or hypertensive encephalopathy;
12. Unstable thrombotic events requiring therapeutic intervention within 6 months prior to screening; Except for infusion set-related thrombosis;
13. Concurrent pulmonary disease leading to severe clinical impairment of respiratory function;
14. Patients with active central nervous system metastases;
15. Patients with large serosal effusions, or symptomatic serosal effusions, or poorly controlled serosal effusions;
16. History of allergy to recombinant humanized antibody or human-mouse chimeric antibody or to any excipient component of the experimental drug;
17. Prior organ transplantation or allogeneic hematopoietic stem cell transplantation;
18. Positive human immunodeficiency virus antibody, active tuberculosis, active hepatitis B virus infection, or active hepatitis C virus infection;
19. Severe infection within 4 weeks prior to first dose of study drug; Lung infection or active lung inflammation within 4 weeks;
20. Have participated in another clinical trial within 4 weeks prior to the first dose;
21. Have a history of psychotropic substance abuse and cannot be abstained from or have a history of severe neurological or psychiatric disorders;
22. Imaging examination showed that the tumor had invaded or encapsulated the large blood vessels in the chest;
23. Severe and non-healing wounds, ulcers, or fractures within 4 weeks prior to signing the informed policy;
24. Clinically significant bleeding or obvious bleeding tendency within 4 weeks prior to signing the informed policy;
25. Subjects who are scheduled to receive or receive a live vaccine within 28 days prior to the first dose;
26. Other conditions that the investigator considers unsuitable to participate in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 24 months
  Objective response rate (ORR) is defined as the number of CR and PR in the treatment and control groups divided by the number of that group in the full analysis set (FAS).
Recommended Phase II Dose (RP2D) | Up to approximately 24 months
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of BL-B01D1.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 24 months
  Progression-free survival (PFS) as assessed by BIRC is defined as the time between the date subjects are randomized and the first observation of disease progression (based on BICR's image-based assessment) or death.
Disease Control Rate (DCR) | Up to approximately 24 months
  Disease Control Rate (DCR) : Percentage of all randomized subjects who rated the best overall response (BOR) as complete response (CR), partial response (PR), and disease stabilization (SD) according to RECIST 1.1 criteria.
Duration of Response (DOR) | Up to approximately 24 months
  Duration of Response (DOR) : defined as the period from the date when tumor response is first recorded to the date when objective tumor progression is first recorded or the date of death.
Treatment Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-B01D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-B01D1.

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, PHD, Principal Investigator — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China